CLINICAL TRIAL: NCT03162991
Title: The Effect of a 12-Week Aerobic Treadmill Exercise on Markers of Glucose Metabolism
Brief Title: Aerobic Treadmill Exercise And Metabolism
Acronym: The A-TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Joshua Sparks, PhD Candidate; Graduate/Research Assistant, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00067271
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Metabolism Disorder, Glucose; Physical Activity; Sedentary Lifestyle
MeSH Terms: conditions — Glucose Metabolism Disorders; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 12-Week Aerobic Exercise Intervention (Experimental)
  Interventions: Other: Aerobic Exercise Intervention
- 12-Week Control Period (No Intervention)

INTERVENTIONS:
Other: Aerobic Exercise Intervention — Aerobic Exercise Intervention- 12-weeks, exercise 3 non-consecutive days/week for ~30-55 minutes per exercise session.
  Arms: 12-Week Aerobic Exercise Intervention

SUMMARY:
Overview- In this study, overweight or obese, sedentary participants (age=35-55 years, n=20) will be randomized to a 12-week control period or an aerobic exercise intervention. Those randomized into the control group will then complete the exercise intervention subsequently. The planned energy expenditure per week of exercise will be 10-12 kilocalories per kilogram of body weight per week. Participants will complete three non-consecutive exercise sessions per week. Body weight, resting metabolic rate via indirect calorimetry, peak oxygen consumption (VO2peak) through graded exercise testing, fasting blood samples, CGM, sleep and dietary habits via self-report, and physical activity monitoring will be completed at prior to and following the aerobic exercise intervention.

DETAILED DESCRIPTION:
Pre-screening- potential participants interested in participating in the proposed research study will be required to perform a pre-screening to assess eligibility. Interested participants will e-mail the research team at TheATEAMstudy@gmail.com and will be contacted by one of the research team members via telephone to discuss the basics of the study and, if the participant is interested, schedule them for an orientation session.

Orientation- following signature of the informed consent by both the participant and the person who obtained the informed consent, a demographics questionnaire and medical history questionnaire will be administered to assess overall health. Following acquisition of the participant's medical history questionnaire, height and weight, will be measured, and from this BMI will be calculated. If the participant is eligible following testing and measurements at orientation, they will be scheduled for a series of baseline visits.

Baseline visits- baseline visit testing will consist of three visits.

At baseline visit 1, participants will come in and have the CGM device placed. For the CGM, a Dexcom G4 Platinum Professional monitor (Dexcom Company, San Diego, CA) will be used. This particular monitor has been approved by the US Food and Drug Administration for use up to 7 consecutive days. This device has a small implantable catheter that will be placed ~2cm to participant preferred side of the umbilicus, a transmitter, and a receiver. This device collects interstitial fluid glucose concentrations every 5 minutes, 24-hours a day, for 7 days. Alongside the CGM for monitoring of blood glucose, each participant will be required to handle a standard glucometer that employs lancets for finger sticks to gain a quick and simple measurement 2 times/day to ensure that there is no drift in the CGM readings. During this visit an actigraph monitor (wGT3X+, Actigraph, LLC, Pensacola, FL) will be placed on the participant's non-dominant or preferred wrist. This Actigraph wGT3X+ monitor is a device that measures activity patterns in an XYZ-directional pathway. It will be worn for 7 consecutive days concurrently with the CGM to aid in the establishment of wake time. A sleep diary will be utilized to aid in the determination of self-report sleep duration, which will include time in bed, sleep time, wake time, and time out of bed. By utilizing a sleep diary in combination with the actigraph monitor, it will allow for ease of interpretation when analyzing the actigraph monitor raw data by providing an estimate as to what sleep/wake time may be. Self-report food intake will be completed via MyFitnessPal (Under Armour™ Connected Fitness, Baltimore, MD), or a standard food diary if necessary, for not only types of food consumed to assess for the effects of meal content, but also time of consumption to assess postprandial blood glucose concentrations for 7 consecutive days. Following this, participants will be scheduled for baseline visit 2.

At baseline visit 2, ~12-24-hours post-baseline visit 1, following a 12-hour fast a 30-minute resting metabolic rate (RMR) test followed by a fasting blood draw and subsequent 120-minute OGTT will be completed. A 30-minute RMR test will be performed to measure oxygen consumption and energy expenditure at rest. For the RMR testing, a Parvo Medics TrueOne 2400 unit (Parvo Medics TrueOne 2400, Salt Lake City, UT), which will be calibrated each time being used, will be utilized. Each participant will have a clear, plastic hood placed over their head while they lay flat on their back resting, without falling asleep for ~30 minutes in a quiet, dimly lit room. After the 30-minute RMR, a fasting blood draw will take place and blood samples will be aliquoted and frozen in a standard VWR -80oC freezer until all blood samples are collected. Participants will then consume a standard 75 gram glucose drink and perform a 2-hour OGTT. Glucose concentration during OGTT will be collected by the CGM device and time points pre-, and 30-,60-,90-, and 120-minutes post-consumption will be used for analysis. Participants will be asked to be as sedentary as possible during this time period as to not disturb the natural uptake and/or clearance of blood glucose that occurs at rest. Upon completion of these tests participants will be scheduled for their baseline visit day 3, ~5-6 days post-baseline visit day 2. During this time period participants will be informed to maintain their normal daily life patterns and to continue to monitor their diet and sleep up until baseline visit 3.

On baseline visit 3, a graded maximal exercise test will be completed. A ramped treadmill test will be performed to assess peak oxygen consumption (VO2peak) through breath-by-breath analysis. The ramped treadmill test protocol will increase speed and incline every 30-seconds until each participant has reached volitional fatigue while simultaneously achieving VO2peak. The same Parvo Medics TrueOne 2400 unit that was utilized for RMR testing will be used for maximal graded exercise testing; however, instead of a hood over the participant's head, a fitted mouth piece will be employed. During the maximal graded exercise test, participants will also be monitored by 12-lead ECG which will be recorded by a Quinton Q-Stress System (Mortara Instrument, Milwaukee, WI) and analyzed primarily by the PI (Joshua R. Sparks) who has been trained and worked in medical situations where this was his primary responsibility. Graded maximal exercise tests will be performed on the Quinton Q-Stress TM65 treadmill. Other trained personnel will be on-site to aid in monitoring each participants exercise blood pressure and rating of perceived exertion (RPE) and will be recorded every two minutes into each stage to make sure no adverse events may be occurring. VO2peak was established through observation of at least two of the following criteria: highest oxygen consumption achieved prior to plateau in oxygen uptake and heart rate with increased work rate, a respiratory exchange ratio ≥ 1.15, a rating of perceived exertion ≥ 17, or achievement of age predicted maximal heart rate using the equation: 220-age. Upon completion of the graded maximal exercise tests, participants will be instructed as to the next stage of the study. Half of the 20 participants (n=10) will be randomized into a 12-week observational control period which precedes the aerobic exercise intervention, while the remainder will immediately begin their aerobic exercise intervention.

The participants that are randomized into the control period will be asked to maintain normal daily activities and will be requested to attend a session once a week for weekly weigh-ins as to observe any fluctuations in weight that may occur over the 12-week control period. Upon completion of the 12-week control period, participants randomized into the control group will undergo pre-intervention testing, which will be designed in the same fashion as baseline testing. Upon completion of the pre-intervention testing, participants will begin their 12-week aerobic exercise intervention.

The 12-week aerobic exercise intervention is designed to elicit physiological changes that occur when currently sedentary, overweight or obese adult begins to become more physically active. Participants will be scheduled to come to the CERC on 3 non-consecutive days per week and exercise to elicit a 10-12 kcal per kilogram of body weight per week energy expenditure while walking at 50-55% Heart Rate Reserve (HRR). Participants will be offered either a morning or an afternoon training session. Which training sessions they choose (morning/afternoon) will be recorded. At each exercise session, prior to beginning their session, body weight, as well as resting heart rate and blood pressure will be recorded. Each session will be supervised by trained personnel. During the exercise session, heart rate will be recorded every five minutes and blood pressure at the mid-way point of the session. Immediately post-exercise heart rate and blood pressure, as well as following a 2-minute rest period will be recorded to verify each participant is recovering without any complications.

Upon completion of the 12-week aerobic exercise intervention, post-intervention testing will take place in the same design as baseline and pre-intervention testing.

ELIGIBILITY:
Inclusion Criteria:

1. be age 35-55 years of age,
2. have 25≤body mass index (BMI)≤40 kg/m2,
3. be weight stable (±2%) during the previous 3 months,
4. have ˂120 minutes of resistance or endurance exercise per week during the previous 3 months, and
5. for females, be eumenorrheic, or post-menopausal for ≥1 year.

Exclusion Criteria:

1. self-reported medical conditions (e.g. diabetes), cardiovascular diseases, chronic or recurrent respiratory conditions (e.g. uncontrolled asthma or chronic obstructive pulmonary disease), active cancer, and eating, or neurological disorders,
2. medications that affect metabolism (e.g. thyroid medications, statins),
3. psychological issues, including but not limited to untreated depression and attention deficit disorder,
4. excessive caffeine use (>500 mg/day),
5. smoking during the past year,
6. pregnant or lactating females,
7. unwillingness to provide informed consent.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Continuous Glucose Monitoring | 3-6 months
  Fasting, Postprandial, and Matched Time Point Glucose Measurements
Glucose Regulatory Hormones | 3-6 months
  Fasting blood concentrations of Glucose Regulatory Hormones

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Research Center, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No